CLINICAL TRIAL: NCT04662190
Title: Eficàcia i Seguretat de la descompressió orbitària en Orbitopatia distiroïdal Utilitzant Models Individualitzats d'impressió 3D Per la planificació i simulació de la Cirurgia.
Brief Title: Evaluation of the Efficacy and Safety of 3D Printing for Orbital Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Collaborators: Societat Catalana d'Oftalmologia (Unknown)
Responsible Party: Principal Investigator, Eduard Pedemonte-Sarrias, Ophthalmologist, MD, PhD, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI 20-16
Record Dates: First submitted 2020-12-06; First posted 2020-12-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Associated Ophthalmopathy; Surgical Procedure, Unspecified
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control grup (Active Comparator): Conventional surgery.
  Interventions: Procedure: Standard surgery
- Intervention group (Experimental): Surgery planned, simulated and guided by 3D printing.
  Interventions: Device: 3D printing model/guide.

INTERVENTIONS:
Device: 3D printing model/guide. — Orbital decompression surgery will be previously planned and simulated using 3D-printed individualized models. In the operating room, surgery will be assisted with 3D-printed individualized guides.
  Arms: Intervention group
Procedure: Standard surgery — Orbital decompression surgery will be previously planned and simulated using the actual standard methods.
  Arms: Control grup

SUMMARY:
This is a multicentric, randomized, single-blinded clinical trial to evaluate the efficacy and safety of 3D printing for the planification and simulation of orbital decompression surgery for thyroid-associated orbitopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inactive thyroid-associated orbitopathy requiring bilateral orbital decompression (moderate-severe in EUGOGO classification).
* Volunteers older than 18 years old.
* Ability to read.
* Acceptation to participate and signature of informed consent.

Exclusion Criteria:

* Younger than 18 years old.
* Previous orbital surgery.
* Any coexisting disease preventing follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative complications | 6 months
  Intraoperative complications
Postoperative complications | 6 months
  Postoperative complications
Exophthalmos | 6 months
  Exophthalmos measured in millimeters
Diplopia | 6 months
  Diplopia correction

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Pedemonte-Sarrias, Md, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (1):
- Eduard Pedemonte Sarrias, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No